CLINICAL TRIAL: NCT06460480
Title: Evaluation of Survival Outcomes After Cardiac Arrest by Monitoring Electroencephalogram, Cerebral Oximetry and Serum Biomarkers
Brief Title: Monitoring After Cardiac Arrest: Electroencephalogram and Cerebral Oximetry in Predicting Outcome
Status: Completed | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 159-2023
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-06

CONDITIONS: Cardiac Arrest; EEG With Periodic Abnormalities; Hypoxic-Ischemic Encephalopathy
Keywords: post-cardiac arrest; electroencephalogram; cerebral oxymetry; biomarkers; brain injury
MeSH Terms: conditions — Heart Arrest; Hypoxia-Ischemia, Brain; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples Without DNA — 2 ml blood samples will be collected during routine intensive care sampling, centrifuged, and gathered to study serum biomarkers of NSE, NRGN, and TREM-2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Because of its high incidence, it is essential to determine the neurological prognosis after cardiac arrest. However, there is not much information to guide post-cardiac arrest care. Also, dynamic monitoring of the state of the brain can help provide information about the patient's prognosis other than previously described serum biomarkers. Therefore, the researchers will monitor postcardiac arrest patients in the intensive care unit for 48 hours by electroencephalogram and cerebral oximetry and collect blood samples for serum biomarkers: neuron-specific enolase (NSE), human neurogranin (NRGN) and human trigger receptor expressed on myeloid cells (TREM-2), which are associated with neuronal damage. And investigate the relation of these data to mortality.

DETAILED DESCRIPTION:
After cardiac resuscitation and intubation, the patient will be followed up with electroencephalogram-based monitoring and cerebral oximetry in the ICU for 48 hours. As standard, post-CPR patients will be sedated with midazolam (0.02- 0.1 mg/kg/s) and remifentanil (0.25- 0.5 mcq/kg/min) for 24 hours.

Brain function measurements will be recorded under sedation for the first 24 hours and without sedation for the second 24 hours. The values recorded were suppression ratio, suppression time, patient state index, oxyhemoglobin and deoxyhemoglobin, and regional oxygen saturation. After 24 hours, a 2 ml blood sample will be taken for biomarkers (NSE, NRGN, TREM-2). Patient survival will be followed up for seven days and 28 days.

The demographic data of the patients (age, gender, body mass index, ASA scores, comorbidities, history of previous operations), blood pressure, heart rate and SpO2, CPR duration, the reason for arrest(4H/4T), and inotropic-vasopressor support before and after arrest will be recorded; GCS, APACHE-2, and SOFA scores will be recorded when the patient is first admitted to the intensive care unit and at the time of cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* experienced cardiac arrest
* permanent spontaneous circulation is maintained for at least 48 hours after CPR
* immediate intensive care follow-up after cardiac resuscitation

Exclusion Criteria:

* • Patients under 18 years of age

  * Presence of previously known neurological disease (cerebral palsy, neurodegenerative disease, encephalitis, etc.)
  * Immunosuppressive patients due to previously known hematological malignancy or solid tumor
  * Patients with a history of head trauma
  * Patients with cardiac arrest within 48 hours after spontaneous circulation is established
  * Patients sedated for more than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older who have experienced cardiac arrest and whose permanent spontaneous circulation is maintained for at least 48 hours after CPR
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
early mortality | from the first day of intensive care admission after cardiac resuscitation until seven days
  the status of the patient as exitus or alive within seven days post cardiac arrest
late mortality | from the first day of intensive care admission after cardiac resuscitation until twenty eight days
  the status of the patient as exitus or alive within twenty eight days post cardiac arrest

SECONDARY OUTCOMES:
supression ratio | from the first hour of intensive care admission until 48 hour
  supression ratio is analyzed from the electroencephalogram monitorization as highest value during time frame
oxyhemoglobin deoxyhemoglobin ratio | from the first hour of intensive care admission until 48 hour
  oxyhemoglobin deoxyhemoglobin ratio is a calculated value on the cerebral oximetry monitorization and recorded as the highest deoxyhemoglobine and lowest oxyhemoglobine values
serum biomarkers | post-cardiac arrest 24th hour
  serum biomarkers as NSE, NRGN, TREM2 will be studied in the blood sample at 24 th hour of post cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Berna Caliskan, MD, Study Director — Haseki Training and Research Hospital Anesthesiology and Reanimation Department; Muhammet Ali Gök, Principal Investigator — Haseki Training and Research Hospital Anesthesiology and Reanimation Department
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Seify M, Shata MO, Salaheldin S, Bawady S, Rezk AR. Evaluation of Serum Biomarkers and Electroencephalogram to Determine Survival Outcomes in Pediatric Post-Cardiac-Arrest Patients. Children (Basel). 2023 Jan 18;10(2):180. doi: 10.3390/children10020180. PMID 36832309
- [Background] Calderone A, Jarry S, Couture EJ, Brassard P, Beaubien-Souligny W, Momeni M, Liszkowski M, Lamarche Y, Shaaban-Ali M, Matta B, Rochon A, Lebon JS, Ayoub C, Martins MR, Courbe A, Deschamps A, Denault AY. Early Detection and Correction of Cerebral Desaturation With Noninvasive Oxy-Hemoglobin, Deoxy-Hemoglobin, and Total Hemoglobin in Cardiac Surgery: A Case Series. Anesth Analg. 2022 Dec 1;135(6):1304-1314. doi: 10.1213/ANE.0000000000006155. Epub 2022 Nov 16. PMID 36097147
- [Background] Dilmen OK, Meco BC, Evered LA, Radtke FM. Postoperative neurocognitive disorders: A clinical guide. J Clin Anesth. 2024 Feb;92:111320. doi: 10.1016/j.jclinane.2023.111320. Epub 2023 Nov 8. PMID 37944401